CLINICAL TRIAL: NCT06134960
Title: A Single-center, Open-label, Single-arm Clinical Study of the Safety and Efficacy of KD-496 CAR-T Therapy in Advanced NKG2DL+/CLDN18.2+ Solid Tumors
Brief Title: NKG2D/CLDN18.21 CAR-T(KD-496) in the Treatment of Advanced NKG2DL+/CLDN18.2+ Solid Tumor
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: KAEDI (Other)
Responsible Party: Principal Investigator, Shen Lin, Shen Lin, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD-496-01
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer; Pancreatic Cancer; Solid Tumor
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KD-496 cell infusion (Experimental)
  Interventions: Biological: KD-496

INTERVENTIONS:
Biological: KD-496 — Autologous genetically modified anti-NKG2DL/CLDN18.2 CAR transduced T cells

SUMMARY:
This is a Phase 1, single-arm, single-center, open-label study to evaluate the safety and effectiveness of NKG2D/CLDN18.2-based CAR-T cells infusion in the treatment of advanced NKG2DL+/CLDN18.2+ solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand the study and voluntarily sign informed consent；
2. Age 18 to 75 years old (including 75 years old), male and female；
3. Patients diagnosed with advanced solid tumors by histopathology or cytology and failed at least 2 prior lines treatment; preferentially enrolled in gastric cancer, pancreatic cancer, etc. Standard treatment recommendations refer to the latest version of the National Comprehensive Cancer Network (NCCN) guidelines or the Chinese Society of Clinical Oncology (CSCO) guidelines；
4. Immunohistochemistry confirmed that NKG2DL/CLDN18.2 was positive (the sum of NKG2DL and CLDN18.2 positive scores ≥5 according to the principle of positive comprehensive score 0~12 points).Tissue specimens for IHC testing must be obtained within 1 year prior to registration for screening or, if not available, new tissue samples must be obtained from a recently obtained surgery or diagnostic biopsy；
5. Subjects must have measurable lesions as defined by the RECIST v1.1 standard;
6. ECOG physical status score 0 to 1;
7. Estimated life expectancy ≥ 3 months;
8. Subjects must have adequate peripheral venous access for peripheral blood mononuclear cell (PBMC) collection;
9. Subjects must meet the following conditions prior to screening precondition. If any of the laboratory tests are abnormal, they can be reviewed within 1 week. If the following conditions are still not met, the screening fails:

1)Absolute neutrophil count ≥1.5×10^9/L, platelets ≥90×10^9/L, hemoglobin ≥90 g/L (no blood transfusion or erythropoietin within 14 days) 2)Coagulation parameters: INR≤1.5 times upper limit of normal (ULN), APTT≤1.5 ULN; 3)Liver function: total bilirubin ≤1.5 ULN; Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 ULN; 4)Renal function: creatinine ≤1.5 ULN or creatinine clearance ≥60ml/min (Cockcroft and Gault formula); 5)Lung function: SaO2≥92%; 6)Cardiac function: Cardiac ejection fraction (LVEF) ≥50% detected by echocardiography or MUGA 1 month before enrollment; 10.Male and female participants of reproductive age agreed to use an approved contraceptive method (e.g., contraceptive pill, barrier device, IUD) for the duration of the study until at least 12 months after the last dose of infusion and two consecutive PCR tests found no CAR T cells.

Exclusion Criteria:

1. Serologically positive for HIV or treponema pallidum, or active hepatitis B (HBV DNA ≥500 IU/mL) or hepatitis C (anti-HCV positive with HCV RNA above the lower limit of assay detection)
2. Any active infection that can't be controlled
3. Patients have autoimmune diseases, have undergone organ transplantation or allogeneic hematopoietic stem cell transplantation, and require long-term systemic glucocorticoid (local use allowed) or other immunosuppressive therapy;
4. History of severe heart disease, including poorly controlled hypertension (SBP >160mmHg and/or DBP >90mmHg), and any of the following conditions that have occurred in the past 6 months: prolonged QT interval syndrome, ECG shows QTc interval >470mSEC, congestive heart failure (New York Heart Association grade ≥ III), cardiac angioplasty and stenting, myocardial infarction, unstable angina, severe arrhythmia, or other heart disease assessed by the investigator as unsuitable for enrollment;
5. Brain metastases with clinical symptoms, except for patients who are stable and asymptomatic lasting at least 14 days after radiotherapy or surgery;
6. Other central nervous system disorders assessed by the investigator to affect the trial: such as seizures, cerebral ischemia/bleeding, dementia, cerebellar diseases, or diseases affecting the central nervous system;
7. Complicated with hematologic malignancies or other primary malignant solid tumors, except for the following cases: 1) patients with cervical cancer or breast cancer in situ with no evidence of disease for more than 3 years after radical treatment; 2) Patients who have successfully received definitive in situ tumor resection without evidence of disease for ≥5 years;
8. Patients with unstable or active peptic ulcer or gastrointestinal bleeding;
9. Received chemotherapy, molecular targeted therapy, interventional therapy, or other antitumor therapy within 3 weeks before apheresis;
10. Patients have received treatment with genetically modified T cells (including CAR-T, TCR-T) or other immune cell therapy previously;
11. Female subjects who are pregnant or breastfeeding;
12. Patients with AEs induced by previous anti-tumor treatment that have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) ≤1, except for alopecia;
13. Received any live vaccine within 2 weeks prior to enrollment;
14. Patients are allergic to precondition drugs (including not limited to fludarabine, cyclophosphamide), allergic to KD-496 injection ingredients (dimethyl sulfoxide, human blood albumin), or have a history of severe allergies (such as anaphylactic shock);
15. Other conditions that investigators considered unsuitable for inclusion;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-16 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | 3 months after infusion
  Incidence of Treatment Related AEs, AEs of special interest and serious adverse events (SAEs)
Dose-limiting toxicity (DLT) rate | 1 month after single infusion
  A drug-related toxicity during treatment with the drug, the severity of which is clinically unacceptable, limiting the further escalation of drug dose.

SECONDARY OUTCOMES:
Objective response rate(ORR) | Up to 1 year after infusion
  objective tumor response rate will be calculated for patients with measurable disease per RECIST 1.1
Duration of Response | Up to 18 months
  Duration of time from first response to progression of disease as determined by investigator
Disease Control Rate | Up to 18 months
  Percentage of patients evaluated as CR and PR determined by investigator
CAR positive T cells in patients | Up to 6 months after infusin
  The time of CAR-T cell reach the peak and turn back to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Professor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No